CLINICAL TRIAL: NCT05759832
Title: Modified Nasal High-flow Oxygen Therapy for Acute Respiratory Failure Patients Undergoing Flexible Bronchoscopy
Brief Title: Modified HFNC Therapy for ARF Patients Undergoing Flexible Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Rui Wang, Attending doctors, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KE-17; PX2023010 (Other Grant/Funding Number: Beijing Hospitals Authority)
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Hypoxemic Respiratory Failure; High-flow Nasal Cannula Oxygen
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified HFNC oxygen therapy group (Experimental)
  Interventions: Device: Modified HFNC oxygen therapy
- Standard oxygen therapy (Other): Non-rebreathing reservoir mask
  Interventions: Device: Non-rebreathing reservoir mask

INTERVENTIONS:
Device: Modified HFNC oxygen therapy — In the modified HFNC group, high-flow devices (AIRVOTM 2; Fisher & Paykel Healthcare, Auckland, New Zealand) were utilized for respiratory support. The nasal cannula used was a modified single nasal cannula.
  Arms: Modified HFNC oxygen therapy group
Device: Non-rebreathing reservoir mask — In the non-rebreathing reservoir mask group, oxygen was delivered via a non-rebreathing reservoir mask during bronchoscopy. The oxygen flow was set to achieve a saturation of pulse oxygen > 90%.
  Arms: Standard oxygen therapy

SUMMARY:
Acute respiratory failure (AFR) is a serious condition that requires prompt and appropriate intervention to prevent further deterioration and improve outcomes. Bronchoscopy is a commonly used diagnostic and therapeutic procedure in patients with respiratory failure. However, traditional low-flow oxygen supplementation during bronchoscopy may not provide adequate oxygenation and ventilation, leading to complications and worsening of the patient's condition.

High-flow nasal cannula therapy has improved oxygenation and ventilation in critically ill patients, making it a promising alternative to traditional oxygen supplementation during bronchoscopy. The bronchoscope is passed through the nose during all procedures in our center. HFNC oxygen therapy is applied to both nostrils. The bronchoscope occupies one of the nares receiving oxygen therapy during bronchoscopy. As a result, the application of HFNC needs to be optimized. Therefore, the investigators designed a modified HFNC with a single cannula. However, limited data exist on the safety and efficacy of modified HFNC therapy in patients with respiratory failure undergoing bronchoscopy.

Therefore, the aim of this study is to evaluate the impact of modified HFNC therapy on the outcomes of undergoing bronchoscopy in patients with ARF. The findings of this study will contribute to understanding the role of modified HFNC therapy in managing ARF and inform clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Respiratory failure defined as a ratio of the partial pressure of arterial oxygen to the fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg;
3. Clinical indication for FB to diagnose or treat pulmonary disease.

Exclusion Criteria:

1. Pre-existing endotracheal intubation or tracheostomy;
2. Required immediate endotracheal intubation;
3. PaO2/FiO2 <150 mm Hg;
4. Platelet count <60 × 109/L;
5. History of myocardial infarction within the past 6 weeks;
6. Nasopharyngeal obstruction or blockage;
7. Presence of chest skin lesions contraindicating the application of electrical impedance tomography (EIT);
8. Intolerance to HFNC oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Need to increase ventilatory support | Within 24 hours after bronchoscopy
  The primary outcome was the need for respiratory support escalation within 24 hours after FB. Escalation was defined as meeting any of the following criteria:
  1. Escalation to invasive mechanical ventilation (IMV);
  2. Escalation to non-invasive ventilation (NIV);
  3. Escalation to HFNC oxygen therapy;
  4. An increase in support parameters without changing the level of respiratory support: For NIV patients: a >20% increase in inspiratory positive airway pressure (IPAP), expiratory positive airway pressure (EPAP), or fraction of inspired oxygen (FiO2); For HFNO patients: a >20% increase in flow rate or FiO2; For low-flow nasal oxygen (LFNO) therapy patients: a >50% increase in oxygen flow rate.

SECONDARY OUTCOMES:
A hierarchy of escalated respiratory support forms based on clinical severity | Within 24 hours after bronchoscopy
  A hierarchical composite outcome, assessed in a fixed sequence: escalation to IMV, escalation to NIV, escalation to HFNO therapy, and an increase in support parameters without changing the level of respiratory support.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Wang, Dr., Study Director — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (2):
- China (2):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Qinghai University, Xining, Qinghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Background] Del Sorbo L, Ferguson ND. High-Flow Nasal Cannulae or Noninvasive Ventilation for Management of Postoperative Respiratory Failure. JAMA. 2015 Jun 16;313(23):2325-6. doi: 10.1001/jama.2015.5304. No abstract available. PMID 25980431
- [Background] Braunlich J, Beyer D, Mai D, Hammerschmidt S, Seyfarth HJ, Wirtz H. Effects of nasal high flow on ventilation in volunteers, COPD and idiopathic pulmonary fibrosis patients. Respiration. 2013;85(4):319-25. doi: 10.1159/000342027. Epub 2012 Nov 1. PMID 23128844
- [Background] Miller EJ. Hypoxemia during fiberoptic bronchoscopy. Chest. 1979 Jan;75(1):103. doi: 10.1378/chest.75.1.103b. No abstract available. PMID 421510
- [Background] Pirozynski M, Sliwinski P, Radwan L, Zielinski J. Bronchoalveolar lavage: comparison of three commonly used procedures. Respiration. 1991;58(2):72-6. doi: 10.1159/000195900. PMID 1862254
- [Background] Fang WF, Chen YC, Chung YH, Woon WT, Tseng CC, Chang HW, Lin MC. Predictors of oxygen desaturation in patients undergoing diagnostic bronchoscopy. Chang Gung Med J. 2006 May-Jun;29(3):306-12. PMID 16924893
- [Background] Longhini F, Pelaia C, Garofalo E, Bruni A, Placida R, Iaquinta C, Arrighi E, Perri G, Procopio G, Cancelliere A, Rovida S, Marrazzo G, Pelaia G, Navalesi P. High-flow nasal cannula oxygen therapy for outpatients undergoing flexible bronchoscopy: a randomised controlled trial. Thorax. 2022 Jan;77(1):58-64. doi: 10.1136/thoraxjnl-2021-217116. Epub 2021 Apr 29. PMID 33927023
- [Background] Douglas N, Ng I, Nazeem F, Lee K, Mezzavia P, Krieser R, Steinfort D, Irving L, Segal R. A randomised controlled trial comparing high-flow nasal oxygen with standard management for conscious sedation during bronchoscopy. Anaesthesia. 2018 Feb;73(2):169-176. doi: 10.1111/anae.14156. Epub 2017 Nov 24. PMID 29171661
- [Background] Irfan M, Ahmed M, Breen D. Assessment of High Flow Nasal Cannula Oxygenation in Endobronchial Ultrasound Bronchoscopy: A Randomized Controlled Trial. J Bronchology Interv Pulmonol. 2021 Apr 1;28(2):130-137. doi: 10.1097/LBR.0000000000000719. PMID 33105418
- [Background] Ben-Menachem E, McKenzie J, O'Sullivan C, Havryk AP. High-flow Nasal Oxygen Versus Standard Oxygen During Flexible Bronchoscopy in Lung Transplant Patients: A Randomized Controlled Trial. J Bronchology Interv Pulmonol. 2020 Oct;27(4):259-265. doi: 10.1097/LBR.0000000000000670. PMID 32265363
- [Background] Simon M, Braune S, Frings D, Wiontzek AK, Klose H, Kluge S. High-flow nasal cannula oxygen versus non-invasive ventilation in patients with acute hypoxaemic respiratory failure undergoing flexible bronchoscopy--a prospective randomised trial. Crit Care. 2014 Dec 22;18(6):712. doi: 10.1186/s13054-014-0712-9. PMID 25529351
- [Background] Li XY, Tang X, Wang R, Yuan X, Zhao Y, Wang L, Li HC, Chu HW, Li J, Mao WP, Wang YJ, Tian ZH, Liu JH, Luo Q, Sun B, Tong ZH. High-Flow Nasal Cannula for Chronic Obstructive Pulmonary Disease with Acute Compensated Hypercapnic Respiratory Failure: A Randomized, Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Nov 24;15:3051-3061. doi: 10.2147/COPD.S283020. eCollection 2020. PMID 33262584
- [Background] Wang R, Li HC, Li XY, Tang X, Chu HW, Yuan X, Tong ZH, Sun B. Modified high-flow nasal cannula oxygen therapy versus conventional oxygen therapy in patients undergoing bronchoscopy: a randomized clinical trial. BMC Pulm Med. 2021 Nov 14;21(1):367. doi: 10.1186/s12890-021-01744-8. PMID 34775948